CLINICAL TRIAL: NCT07108569
Title: Ability of Physicians to Distinguish Real From Artificial Colon Polyp Images
Acronym: LUTETIA1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022120701
Record Dates: First submitted 2024-08-08; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Colon Polyp; Colonic Adenoma
Keywords: Colonoscopy
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Masking Description: Participant does not know if pesented image is real or artificial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Image assessment (Experimental): Physicians judge whether the random image presented to them is real or artificial
  Interventions: Other: Lutetia

INTERVENTIONS:
Other: Lutetia — Lutetia is an AI-based training plattform

SUMMARY:
Training in endoscopy is essential for the early detection of precursors of colorectal cancer. Up to now, this training has been carried out with image collections of findings and in practice when working on patients.

The investigators want to use artificial intelligence (AI) to better train doctors to recognise these precursors. By using generative AI, the investigators were able to create realistic images that comply with data protection regulations and whose content can be predefined. Parts of the image can also be regenerated so that it is possible to create different precancerous stages in the same place in the image.

In this study the investigators want to identify the ability of physicians to distinguish artificial from real polyp images.

ELIGIBILITY:
Inclusion Criteria:

* Physicians with or without experience in colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Ability to detect artificial images as artificial | 6 months
  The ability to recognise artificial images as being artificial, using an online questionnaire - binary question

SECONDARY OUTCOMES:
Ability to detect real images as real | 6 months
  The ability to recognise real images as being real using an online questionnaire - binary question
Accuracy to correctly classify images | 6 months
  Accuracy to correctly classify images using an online questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hann, MD, Principal Investigator — Wuerzburg University Hospital
Locations (1):
- University hospital Würzburg b, Würzburg, Germany